CLINICAL TRIAL: NCT06918444
Title: Effect of the WARIFA App on User-defined Objectives, Healthy Lifestyles and Management of Type 1 Diabetes: a Pilot Randomised Controlled Trial
Brief Title: Evaluation of the WARIFA App and Its Impact on Healthy Lifestyle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Universitario de Investigaciones Biomédicas y Sanitarias (iUIBS) de la Universidad de Las (Other)
Collaborators: Complejo Hospitalario Universitario Insular Materno Infantil (Other)
Responsible Party: Principal Investigator, Rosa María Sánchez Hernández, MD, PhD, Complejo Hospitalario Universitario Insular Materno Infantil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-330-1
Record Dates: First submitted 2024-10-06; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Lifestyle Intervention; Non Communicable Chronic Diseases; Type 1 Diabetes (T1D)
Keywords: AI (Artificial Intelligence); Mobile app; Lifestyle intervention; Non Communicable Chronic Diseases; Risk Prediction Model; Type 1 Diabetes (T1D)
MeSH Terms: conditions — Noncommunicable Diseases; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use of WARIFA app with artificial intelligence (AI) (Experimental): Participants will use a version of WARIFA app with artificial intelligence and personalized messages.
  Interventions: Device: WARIFA app with AI
- Use of WARIFA app without artificial intelligence (AI) (Placebo Comparator): Participants will use a version of WARIFA app with the same functionalities as the intervention group, but without artificial intelligence and personalized messages.
  Interventions: Device: WARIFA app without AI

INTERVENTIONS:
Device: WARIFA app with AI — Participants will be given access to the WARIFA app on their mobile phones during the study.
  This app will collect activity data as well as questionnaires and diaries. Using this data and artificial intelligence, it will provide participants with personalised information and recommendations about their lifestyle and risk of chronic non-communicable diseases.
  Arms: Use of WARIFA app with artificial intelligence (AI)
Device: WARIFA app without AI — Participants will be given access to the WARIFA app on their cell phones during the study.
  This app will collect activity data, as well as through questionnaires and diaries. With this data, it will give information and general recommendations to the participants related to their lifestyle habits and risks of chronic non-communicable diseases, following the WHO guidelines. This version will not use artificial intelligence or personalized messages.
  Arms: Use of WARIFA app without artificial intelligence (AI)

SUMMARY:
The goal of this study is to assess the effect of the WARIFA app on the adoption of healthy lifestyle behaviours related to Non-communicable diseases (NCDs), as well as in the management of Type 1 Diabetes (T1D). This is done using user-generated data analysis, artificial intelligence (AI) and risk estimation to provide personalised recommendations on lifestyle-related behaviours through a mobile app.

* Primary objective: the objective of this study is to assess the impact of using the WARIFA app on a series of outcomes, related to the promotion of healthy lifestyles and prevention of NCDs, as well as on the management of T1D.
* Secondary objectives: to assess the feasibility of implementation of a complex health app (WARIFA), and to explore which outcomes are more relevant in this context for users.

The study will evaluate the app in two different populations:

* Population 1: Citizens living in Europe of either sex aged > 18 years diagnosed with no more than one NCD (of the following: CVD, any type of cancer, chronic respiratory disease and T2D) and current owners of a smartphone with internet access.
* Population 2: European adult individuals of either sex aged >18 years with T1D currently using multiple daily insulin injections or an insulin pump and current owners of a smartphone with internet access.

The study will be carried out in three centres in three different countries: the Instituto Universitario de Investigaciones Biomédicas y Sanitarias (iUIBS) in Spain, the Norwegian Centre for E-health Research (NSE) in Norway, and in Romania.

Participants in each population will be randomised to an intervention or control arm on a 1:1 ratio:

* Intervention arm: the Warifa app will be used by the participants throughout the study. The app will provide personalised risk estimations and recommendations through user-generated data analysis and artificial intelligence.
* Control arm: The control group will use a Warifa app with the same functionalities than the intervention arm, but without artificial intelligence.

At baseline, information will be collected by questionnaires and a physical examination, including anthropometry and a lipid profile. These measurements will be repeated in 12 weeks and will be compared between the treatment arms.

The study will last 3 months in total, start of recruitment on 10 February 2025, end of study after the last visit of the last participant, on 12 May 2025. Each user will participate in the study for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Common for both population groups:
* Adults over 18 years of age.
* Owners of a smartphone operating with Android and with internet access.
* Group 1: General population:
* Healthy or diagnosed with no more than one NCD (CVD, any type of cancer, T2D or chronic respiratory disease).
* Group 2: T1D:
* Treatment with multiple subcutaneous insulin injections or an insulin pump.
* Users of a continuous glucose monitor.

Exclusion Criteria:

* Common for both groups:
* Pregnancy.
* Mobile device which is incompatible with the WARIFA app (E.g. Apple devices).
* Unable to understand any of the app languages (Spanish, English, Norwegian or Romanian).
* Any reason which precludes follow-up, based on the researcher's criteria.
* Group 1: General population
* People with two or more NCDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-29 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Self-defined goal by the participants | At the end of intervention at 12 weeks
  Degree of achievement of a self-defined goal by the participants (selected among: increase consumption on fruit and vegetables, increase physical activity, reduce alcohol consumption, stop smoking, reduce number of weekly hypoglycaemic episodes, or improve sun protective behaviours).
  It will be measured on a Likert scale, with scores ranging from 1 ('well below expectations') to 10 ('well above expectations').

SECONDARY OUTCOMES:
Frequency of app use | From enrollment to the end of intervention at 12 weeks
  Number of times users access the app (number of times per day). Direct adherence.
Time spent using the app | From enrollment to the end of intervention at 12 weeks
  Time spent using the app (number of hours per day). Direct adherence.
Consistency in data recording | From enrollment to the end of intervention at 12 weeks
  Assessment of the regularity with which users record information related to healthy habits, healthy eating and physical activity. Direct adherence.
ABACUS scale | At the enrollment and the end of intervention at 12 weeks
  The validated App Behaviour Change Scale (ABACUS). Attitudinal/Behavioural Change. The ABACUS scale was designed to measure the potential behavior change of apps. It consists of 21 items grouped into 4 categories: knowledge and information (5 items), goals and planning (3 items), feedback and monitoring (7 items), and actions (6 items). Each item represents a behavior change technique, and its inclusion in the app is rated dichotomously (behavior change technique not included = 0 or included = 1). Higher score means more potential behavioural change of apps.
Changes in eating habits | From enrollment to the end of intervention at 12 weeks
  Assessment of changes in diet quality (changes in consumption of fruits, vegetables, processed foods…). Diary recording of fruit, vegetable, and processed meat consumption will be used. Attitudinal/Behavioural Change.
Changes in physical activity | From enrollment to the end of intervention at 12 weeks
  Data collected through a compatible smartwatch (number of steps) will be recorded. Attitudinal/Behavioural Change.
Reduction in tobacco consumption | From enrollment to the end of intervention at 12 weeks
  Diary records of tobacco consumption will be used (number of cigarettes per day). Attitudinal/Behavioural Change.
Reduction in alcohol consumption | From enrollment to the end of intervention at 12 weeks
  Diary records of alcohol consumption will be used (Number of units of alcoholic beverages per day). Attitudinal/Behavioural Change.
Changes in sun protection behaviour | At the enrollment and the end of intervention at 12 weeks
  sun habits questionnaire score wil be used. Attitudinal/Behavioural Change
Changes in sun protection behaviour | From enrollment to the end of intervention at 12 weeks
  Daily record of sunscreen use. Attitudinal/Behavioural Change
Hypoglycaemic events | From enrollment to the end of intervention at 12 weeks
  The continuous glucose monitor data from participants will be used (number of hypoglycaemic events). Biomedical outcomes
Hypoglycaemic events | From enrollment to the end of intervention at 12 weeks
  Diary records of manually recorded hypoglycaemic events (number of hypoglycaemic events). Biomedical outcomes.
Glycosylated haemoglobin | At the enrollment and the end of intervention at 12 weeks
  Will be measured in venous blood. Unit of measurement: %. Biomedical outcomes.
Glucose Management Indicator | From enrollment to the end of intervention at 12 weeks
  Glucose Management Indicator in the last 14 days. Unit of measurement: %. Biomedical outcome
Average glucose | From enrollment to the end of intervention at 12 weeks
  Average glucose in the last 14 days. Unit of measurement: mg/dl. Biomedical outcomes.
Time in ranges | From enrollment to the end of intervention at 12 weeks
  Times in glucose range for the last 14 days, measured by the participants' glucose sensor. Unit of measurement: %. Biomedical outcomes.
Total cholesterol | At the enrollment and the end of intervention at 12 weeks
  Total cholesterol, measured through a venous blood sample. Unit of measurement: mg/dl. Biomedical outcomes.
HDL cholesterol | At the enrollment and the end of intervention at 12 weeks
  HDL cholesterol, measured through a venous blood sample. Unit of measurement: mg/dl. Biomedical outcomes.
LDL cholesterol | At the enrollment and the end of intervention at 12 weeks
  LDL cholesterol, measured through a venous blood sample. Unit of measurement: mg/dl. Biomedical outcomes.
Non-HDL cholesterol | At the enrollment and the end of intervention at 12 weeks
  Non-HDL cholesterol, measured through a venous blood sample. Unit of measurement: mg/dl. Biomedical outcomes.
Muscle mass. | At the enrollment and the end of intervention at 12 weeks
  Muscle mass. Measured by impedanciometry. Unit of measurement: Kg. Biomedical outcomes.
Fat mass | At the enrollment and the end of intervention at 12 weeks
  Fat mass. Measured by impedanciometry. Unit of measurement: Kg. Biomedical outcomes.
Weight | At the enrollment and the end of intervention at 12 weeks
  Weight of each participant. Unit of measurement: Kg. Biomedical outcomes
Height | At the enrollment
  Height of each participant. Unit of measurement: cm. Biomedical outcomes
Circumference of abdomen. | At the enrollment and the end of intervention at 12 weeks
  Circumference of abdomen. Unit of measurement: cm. Biomedical outcomes
Circumference of the calf | At the enrollment and the end of intervention at 12 weeks
  Circumference of the calf. Unit of measurement: cm. Biomedical outcomes
Dynamometry | At the enrollment and the end of intervention at 12 weeks
  Functional test, using a dynamometer in each participant's hand. Unit of measurement: Kg. Biomedical outcomes
Body fat. | At the enrollment and the end of intervention at 12 weeks
  Measured by plicometer in the posterior region of the upper arm (triceps area). Unit of measurement: mm. Biomedical outcomes.
Chair test 5 repetitions | At the enrollment and the end of intervention at 12 weeks
  Functional test, which measures the time taken to stand up and sit down from a chair 5 times. Unit of measurement: seconds. Biomedical outcomes.
Perceived quality of life | At the enrollment and the end of intervention at 12 weeks
  The EQ-5D questionnaire will be used for the group from the general population. Quality of Life and Wellbeing. Questionnaire with two distinct parts. The first part contains five health dimensions (mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression). For each dimension of the EQ-5D, severity levels are coded: 1 if the answer choice is 'no (I have) problems'; 2 if the answer choice is 'some or moderate problems'; and 3 if the answer choice is 'many problems'. The higher the score, the worse the health dimension.
  The second part of the EQ-5D is a scale from 0 to 100. On this scale, the individual should mark the point that best reflects their assessment of their overall health status, with 0 being the lowest assessment of their health status and 100 being the best.
Perceived quality of life | At the enrollment and the end of intervention at 12 weeks
  The "Vida con Diabetes tipo 1" (ViDa1) questionnaire will be used for the group of individuals with T1D. Quality of Life and Wellbeing.
  The ViDa1 has 34 items that are grouped into 4 different dimensions: interference with life, self-care, well-being and worry about the disease. It is a questionnaire that can be self-administered with a Likert-type response format in which a total score per subscale is obtained.
  Interference with life: (items 1 - 12), self-care (13 - 23), well-being (24 - 29) and worry about illness (30 - 34). Each item is scored from 1 'strongly disagree' to 5 'strongly agree'. For correction, the scores obtained in each subscale are added together. Items 12, 23 and 27 are reversed for correct interpretation.
Acquired knowledge | At the enrollment and the end of intervention at 12 weeks
  Assessment of new knowledge about healthy habits. The European Health Literacy Survey will be used. Knowledge and Attitudes.
  The questionnaire consists of 16 questions that classify the degree of difficulty perceived by the participant in each task or situation as: 1 'very easy', 2 'easy', 3 "difficult", 4 'very difficult' or 5 'don't know/no answer'.
Self-efficacy | At the enrollment and the end of intervention at 12 weeks
  For measuring diabetes self-management behaviours, we will use the Summary of Diabetes Self-Care Activities (SDSCA). Knowledge and Attitudes.
  Is a brief self-report questionnaire of diabetes self-management that includes items assessing the following aspects of the diabetes regimen. It consists of 11 items that addresses different areas of self-care present in people with Diabetes Mellitus, such as diet, physical activity, medication, self-testing of capillary glycaemia and smoking. It presents a response scale from 0 to 7, depending on the number of days that the person has carried out a certain behaviour in the last week. The smoking item has a dichotomous response scale.
  The lower the score, the lower the adherence of the person with MD to favourable self-care behaviours. The questionnaire has no cut-off point, so each item must be assessed individually.
Usability | At the enrollment and the end of intervention at 12 weeks
  Usability scale (SUS) will be used. Satisfaction and feedback.
  The SUS scale is a 10-item questionnaire scored on a 5-point Likert-type scale from 1 (strongly disagree) to 5 (strongly agree). It is arranged to alternate between positive and negative statements to avoid habitual bias from the respondent. The score contribution for the odd items (the positive statements) is the scale position minus 1 and the contribution for the even items (the negative statements) is 5 minus the scale position. The overall score is calculated from the sum of all item scores multiplied by 2.5, with the overall score ranging from 0 to 100. A system with a score above 85 is considered to have excellent usability, whereas a system with a score between 68 and 84 is considered to have good usability.
Usability | At the enrollment and the end of intervention at 12 weeks
  The mHealth App Usability Questionnaire (MAUQ) will be used. Satisfaction and feedback.
  It assesses the ease of use, interface, satisfaction and usefulness of mHealth applications for end users. Consists of 18 items, with 7 response options for each item, ranging from 1 "strongly disagree" to 7 "strongly agree".

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Universitario De Investigaciones Biomédicas y Sanitarias (IUIBS), Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No
The study will be conducted in three European countries, in compliance with both national and European data protection laws.

REFERENCES:
- See also: WARIFA project home page — https://www.warifa.eu/